CLINICAL TRIAL: NCT04213768
Title: LR Resection Versus Plication in Esotropia
Brief Title: Lateral Rectus Resection Versus Lateral Rectus Plication in Patients With Residual Esotropia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamideh Sabbaghi, PhD student, Teacher Assistant, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.SBMU.ORC.REC.1398.022
Record Dates: First submitted 2019-12-18; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Strabismus
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plication (Experimental)
  Interventions: Procedure: Lateral rectus plication
- Resection (Active Comparator)
  Interventions: Procedure: Lateral rectus Resection

INTERVENTIONS:
Procedure: Lateral rectus plication — The technique is the same as resection up to the muscle suturing, in the next step, the sutures is passed through 2 scleral bites at 1 mm anterior to the muscle insertion, then the muscle is folded anteriorly by Stevens muscle hook during tightening and fixing the sutures. At the end, conjunctiva is repaired by Vicryl 8-0.
  Arms: Plication
Procedure: Lateral rectus Resection — Following conjunctiva and tendon capsule incision, lateral rectus is hooked and dissected from its surrounding tissues. Then, the muscle is sutured according to the amount of supposed resection from lateral rectus insertion by Vicryl 6-0 (polyglation 910, coated Vicryl®, Ethicon, Blue Ash, OH). Afterwards, the muscle is cut at 1mm anterior to these sutures and the residual muscle is re-sutured to the sclera at its primary insertion. Finally the conjunctiva is repaired using Vicryl 8-0.
  Arms: Resection

SUMMARY:
In this study, the surgical outcomes of lateral rectus plication and resection techniques on patients with residual esotropia will be compared.

Methods: In this randomized clinical trial, a total of 57 patients with residual esotropia (31 females and 26 males) who were candidate for lateral rectus resection are going to be included and randomized into plication and resection groups. The inclusion criteria will be residual esotropia after uni- or bilateral medial rectus recession, or unilateral recession and resection (R&R). Subjects with a history of prematurity, lack of central fixation, extraocular muscle palsy, systemic, ocular disorders, follow up less than three months will be excluded. A comprehensive ophthalmic examinations are going to be conducted preoperatively and at 1, 3 and 6 months' follow-ups. Surgical success rate will be considered in cases with a postoperative eso- or exotropia ≤10pd.

DETAILED DESCRIPTION:
In this clinical trial study, a total of 57 patients with residual esotropia (31 females and 26 males) who were candidate for lateral rectus resection will be included and randomized into plication (n=27) and resection (n=30) groups.

An informed consent will be obtained from all patients or their parents after explanation of the two techniques and their possible advantages and disadvantages. The study protocol will be approved by the Ethics Committee of Ophthalmic Research Center, Shahid Beheshti University of Medical Sciences, Tehran, Iran and it adheres to tenets of the Declaration of Helsinki.

The inclusion criteria will be the presence of residual esotropia ≥15pd after uni- or bilateral medial rectus recession. Subjects with a history of prematurity, intellectual disability, lack of central fixation (nystagmus, eccentric fixation, retinopathy of prematurity), extraocular muscle palsy, systemic, ocular, and neurological disorders, or follow- up less than three months will be excluded from this study. The surgeon who performed surgeries will not be masked, while the personnel who conducted data gathering and postoperative examinations will be blind to the group assignments.

Visual and Ocular Examinations Comprehensive ophthalmic examination including cyclorefraction (45 minutes after installation of one drop tropicamide 1% and cyclopentolate 1%), best corrected visual acuity (BCVA), extraocular muscle motility (version and duction from -4 to +4) will be performed, the ocular deviation will be measured at both far (6m) and near (33cm) distances using an alternate prism cover test or Krimsky method. A- or V- ocular pattern will be also determined if the difference of deviation was more than 10 or 15pd at 30 degrees between superior and inferior of primary position, respectively. Stereopsis will be measured using a Titmus test. According to the patients' response, stereopsis was also classified in to three groups of central (≤100 sec/arc), peripheral (100 to 3000 sec/arc) and suppression (≥3000). Ocular anterior and posterior segments will be examined using slit lamp and indirect ophthalmoscopy. Eligible patients will be randomly divided to lateral rectus plication (case) and lateral rectus resection (control) groups and the amount of operation will be according to the Park's table in the both groups. In patients with residual esotropia less than 20pd, unilateral lateral rectus recession and in patients with residual esotropia more than 20pd, bilateral lateral rectus recession will be considered. All examinations will be repeated at one, three and six month follow-ups. Surgical success rate will be considered in patients with a postoperative deviation ≤10pd.

ELIGIBILITY:
Inclusion Criteria:

- residual esotropia after any strabismus surgery

Exclusion Criteria:

* Subjects with a history of prematurity
* lack of central fixation
* extraocular muscle palsy
* systemic disorders
* ocular disorders
* follow up less than three months

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative angle of deviation measured by alternative prism cover test based on prism diopter unit | 6 months

SECONDARY OUTCOMES:
Postoperative exodrift | 6 months
  Exodrift can be achieved by the change of the post- and preoperative angle of deviation measured by alternative prism cover test at far distance and recorded based on prism diopter unit.

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Hamideh Sabbaghi, Tehran
  - Islamic Republic of Iran, Tehran

IPD SHARING:
Plan to Share IPD: No